CLINICAL TRIAL: NCT04766944
Title: Incidence and Associated Risk Factors of Augmented Renal Clearance (ARC) in Critically Ill Trauma Patients of 50 Years Old and Above
Brief Title: Incidence and Associated Risk Factors of ARC in the Trauma Critically Ill Older Than 50 Years Old
Status: Withdrawn | Type: Observational
Why Stopped: This study was planned and approved just before the 2020 pandemic - once the pandemic resolved, significant changes occurred in the ICU that prevented doing the study - hence it was withdrawn with no patient ever enrolled
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Marc M. Perreault, Full clinical professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6327
Record Dates: First submitted 2021-02-14; First posted 2021-02-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Augmented Renal Clearance; Critical Illness; Polytrauma; Traumatic Brain Injury
Keywords: Augmented renal clearance; Critical illness; Critical care; Intensive care unit; Trauma; Polytrauma; Traumatic brain injury; Elderly; Middle-aged
MeSH Terms: conditions — Critical Illness; Multiple Trauma; Brain Injuries, Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine collected from a daily 8-hour collection via an indwelling urinary catheter will be used to assess total daily urine volume. Urine samples of 2 ml will be taken and kept in a biomedical laboratory freezer at -80°C to be analyzed in batches every 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill trauma patients of 50 years old and above: Patients of 50 years old and above admitted to the Montreal General Hospital intensive care unit for trauma
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This single-center prospective cohort study conducted at the adult trauma ICU of the Montreal General Hospital (MGH) affiliated with the McGill University Health Centre (MUHC) aims to determine the incidence and associated risk factors of augmented renal clearance (ARC) in critically ill trauma patients of 50 years old and above.

DETAILED DESCRIPTION:
Patients aged 50 years or older admitted to the ICU for traumatic brain injury (TBI) and/or polytrauma between January 2021 and October 2021 will be screened for study enrollment according to inclusion and exclusion criteria.

Research hypothesis :

* Critically ill trauma patients aged 50 years or older admitted to the ICU present an augmented renal clearance;
* A set of factors could predict, to a certain extent, the risk of developing ARC in critically ill trauma patients aged 50 years or older admitted to the ICU.

ARC will be assessed for every patient based on daily 8-hour urine collections started within the first 24 hours of ICU admission and daily serum creatinine concentrations. The first seven days will consist of daily urinary collection while only biweekly samples (days 10 and 14) will be collected for the second week. Since ARC is a time-sensitive event, the use of a deferred consent will allow for urine collection to begin as soon as possible after admission. All other data required for the study (demographic and other clinically relevant data) will be collected retrospectively once consent from surrogate or patient has been obtained. Data will be collected from study enrollment up until one of the following events : 1) Day 14 of ICU stay ; 2) ICU discharge; 3) AKI onset; 4) institution of RRT; 5) Removal of urinary catheter; 6) Withdrawal of informed consent; 7) Death; whichever occurs first.

Data regarding demographic variables including age, gender, anthropometric measurements, admission diagnosis, nature of injuries, comorbidities, and length of stay (LOS) will be obtained through the patient's medical records as well as the clinical information system. Data concerning ventilation and 24-hour fluid balance will be obtained through nursing records. Information regarding drug therapy (e.g., vasopressor and antibiotic use) will be obtained through the MUHC software. The Injury Severity Score (ISS) score will be compiled from the local Trauma Registry, while the Sequential Organ Failure Assessment (SOFA) score will be calculated directly.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU for isolated traumatic brain injury (TBI), polytrauma without TBI or combined polytrauma and TBI
* Expected ICU length of stay of more than 24 hours
* Age of ≥ 50 years old at the time of admission
* Serum creatinine ≤ 120 μmol/L at the time of admission
* Presence of an indwelling urinary catheter
* Consent is obtained from the patient or its surrogate decision-maker within 7 days of ICU admission

Exclusion Criteria:

* History of renal replacement therapy (RRT) (intermittent dialysis or peritoneal dialysis), nephrectomy or renal transplant
* Patient developing acute kidney injury (AKI)
* ICU physician considered patient unsuitable for enrollment due to poor prognosis
* Burn-related trauma
* Patient is admitted > 48 hours post-traumatic event

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 years old or older admitted to the ICU for traumatic brain injury (TBI) and/or polytrauma between January 2021 and October 2021
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of augmented renal clearance in critically ill trauma patients aged 50 years and older | Once a day, up to 14 days
  The incidence of augmented renal clearance is dichotomic: presence or absence of augmented renal clearance defined as a creatinine clearance of ≥ 130 mL/min/m² measured by a daily 8 hour urine collection

SECONDARY OUTCOMES:
To determine demographic and clinical risk factors for ARC in critically ill trauma patients aged 50 years and older | Up to 14 days
  Predictive variables of ARC to be included in the model include: age strata (50-59 years old, 60-69 years old, 70 years old and above; biological gender; type of trauma (TBI, polytrauma without TBI, combined polytrauma and TBI) and severity of trauma (Injury Severity Score (ISS score), Sequential Organ Failure Assessment (SOFA) score, severity of TBI (GSC score at admission).
  Other variables to be included in the model will depend on the number of cases observed with a minimum of 10 cases per variable.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Not at the present time